CLINICAL TRIAL: NCT01880957
Title: Pathophysiology and Treatment of Bipolar Disorder as Assessed by in Vivo Imaging
Brief Title: PET and MRI Brain Imaging of Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The Dana Foundation (Other)
Responsible Party: Principal Investigator, Ramin Parsey, Professor and Chair of the Department of Psychiatry and Director of Positron Emission Tomography (PET) Research, Stony Brook University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-1826-F; 7R01MH090276-03 (NIH)
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Results first posted 2022-06-29 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Bipolar Disorder; Bipolar Depression; Unipolar Depression
Keywords: bipolar disorder; bipolar depression; serotonin transporter; serotonin receptors; binding potential; brain imaging; unipolar depression
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder | interventions — Lithium; Lithium Carbonate; Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lithium (Other): Patients in this condition will receive lithium administered as follows: Day 1, 2 and 3, 300 mg bid; Days 4-7 lithium 300 qam and 600 qhs. Lithium level will be checked as close to Day 7 as possible and titrated to a therapeutic plasma level of 0.8-1.2 mEq/l. Subjects will not undergo lithium monotherapy if they have a documented history of at least two failed trials of lithium of at least 4 weeks duration with therapeutic blood levels for a major depressive episode
  Interventions: Drug: Lithium
- Lamotrigine (Other): Patients who have not respond to adequate prior lithium treatment while depressed, or who refuse lithium, will be given lamotrigine. Lamotrigine will be started at 25 mg bid and increased to 50 mg bid after 2 weeks and again increased to 100 mg bid after an additional 2 weeks.
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lithium
  Other Names: lithium carbonate
  Arms: Lithium
Drug: Lamotrigine
  Other Names: Lamictal
  Arms: Lamotrigine

SUMMARY:
The primary aims of this study are to:

1. Quantify serotonin transporter (5-HTT) binding potential (BP) in vivo in bipolar disorder patients (BPD) during a major depressive episode (MDE).
2. Assess the effect of lithium treatment of bipolar disorder on 5-HTT.
3. Assess the effect of lithium treatment of bipolar disorder on 5-HT1A BP.
4. Assess the effect of lamotrigine treatment of bipolar disorder on 5-HTT and 5-HT1A BP.
5. Assess the effect of lithium treatment of unipolar depression on 5-HTT BP.

DETAILED DESCRIPTION:
PET and MRI imaging will be used to investigate the aims described above in patients who have bipolar disorder or unipolar depression and are currently experiencing a depressive episode. Both healthy controls and depressed participants with bipolar disorder or unipolar depression will be recruited. Patients who are on medication before enrolling in the study will have a three week washout. At baseline, healthy controls and patients will have an MRI consisting of both structural and functional sequences. Psychological measures will also be obtained at baseline. Within one week of the MRI, both patients and healthy controls will have one CUMI and one DASB PET scan.

Following the baseline PET scans, patient participants will begin medication treatment with either lithium or lamotrigine, based on the clinical judgement of the treating psychiatrist. Psychological measures will be obtained every 2 weeks. After 6 weeks of medication treatment at a therapeutic dose, patients will be assessed for remission (defined as a 50% decrease in the HDRS score from baseline). If this criteria is met, patient participants will then have follow-up PET scans (one CUMI and one DASB). If this criteria is not met, the patient will be switched to the other medication under study and will be reevaluated after an additional 4 weeks of medication treatment. Patients who still do not demonstrate a 50% decrease in their HDRS will be considered non-responders and will have repeat CUMI and DASB scans.

ELIGIBILITY:
PATIENTS

BIPOLAR

Inclusion Criteria:

* Bipolar patients suffering from a major depressive episode currently or recently (in the month prior to scanning). Patients on psychiatric medication will have failed their current regimen for the treatment of their depression: they will meet criteria for depression, be seeking treatment for it, and have been on an adequate dose of antidepressant or mood stabilizer (as defined by the Antidepressant Treatment Form-see Oquendo et al., 2003) for 4 weeks or more.
* Of sufficient severity to score at least 15 on the first 17 items of the Hamilton Depression Rating Scale or a score of 10 to 14 on the first 17 items of the Hamilton Depression Scale in conjunction with a score of at least 29 on the Beck Depression Inventory.
* Age range 18-65 years.
* Off all psychotropic and other types of drugs likely to interact with serotonin transporters and 5-HT1A receptors for at least 21 days. Allowed short-acting benzodiazepines for distressing anxiety or insomnia (up to 24 hours prior to each PET scan). Patients will be off neuroleptics for 3 weeks and off fluoxetine for 6 weeks prior to study. Off serotonin depleting drugs such as reserpine for 3 months. Patient will also be off anti-coagulant/anti-platelet treatment such as coumadin, with the exception of aspirin for 10 days.
* Willing to travel for PET scanning

Exclusion Criteria:

* Other major psychiatric disorders such as schizophrenia, schizoaffective illness; current drug or alcohol abuse (within past 2 months), or drug or alcohol dependence <6mos ago; anorexia nervosa or bulimia nervosa in the past year; IV drug use or ecstasy use more than two times.
* A first-degree family history of schizophrenia if the subject is less than 33 years old (mean age of onset for schizophrenia plus two standard deviations).
* Significant active physical illness particularly those that may affect the brain or serotonergic system including blood dyscrasias lymphomas, hypersplenism, endocrinopathies, renal failure or chronic obstructive lung disease, autonomic neuropathies, peripheral vascular disease, diabetes, low hemoglobin and malignancy, significant anemic disease or blood loss and the lab parameters platelet count < 80,000.
* Lacks capacity to consent.
* Actively suicidal-begins expressing a plan for suicide during the washout phase or develop suicidal ideation that warrants admission or requires medication or treatment intervention.
* Electroconvulsive therapy (ECT) within the past 6 months.
* Pregnancy, currently lactating; planning to conceive during the course of study participation or abortion in the past two months.
* Metal implants, pacemaker or metal prostheses or orthodontic appliances, the presence of shrapnel
* Current, past or anticipated exposure to radiation, that may include: being badged for radiation exposure in the workplace, participation in nuclear medicine procedures, including research protocols in the last year.
* A neurological disease or loss of consciousness for more than a few minutes
* Medicinal Patch (participants will be asked to remove before MRI)
* Patients who are responding satisfactorily to psychiatric medications, because they will not be washed-out for purposes of this study
* A documented history of a lack of response to a trial of adequate dose and duration of both lithium and lamotrigine defined as minimal clinical response to lamotrigine 200 mgs for at least 4 weeks or lithium serum levels of at least 0.8 (or dose >= 900 mgs) for at least 4 weeks.
* Patient is unlikely to be able to tolerate medication washout
* Claustrophobia
* Blood donation within 8 weeks of the start of the study.
* History of bleeding disorder or are currently taking anticoagulants.

UNIPOLAR

Inclusion:

* Unipolar patients suffering from a major depressive episode currently or recently (in the month prior to scanning). Patients on psychiatric medication will have failed their current regimen for the treatment of their depression: they will meet criteria for depression, be seeking treatment for it, and have been on an adequate dose of antidepressant or mood stabilizer (as defined by the Antidepressant Treatment Form-see Oquendo et al., 2003) for 4 weeks or more.
* Of sufficient severity to score at least 15 on the first 17 items of the Hamilton Depression Rating Scale or a score of 10 to 14 on the first 17 items of the Hamilton Depression Scale in conjunction with a score of at least 29 on the Beck Depression Inventory.
* Age range 18-65 years.
* Off all psychotropic and other types of drugs likely to interact with serotonin transporters and 5-HT1A receptors for at least 21 days. Allowed short-acting benzodiazepines for distressing anxiety or insomnia (up to 24 hours prior to each PET scan). Patients will be off neuroleptics for 3 weeks and off fluoxetine for 6 weeks prior to study. Off serotonin depleting drugs such as reserpine for 3 months. Patient will also be off anti-coagulant/anti-platelet treatment such as coumadin, with the exception of aspirin for 10 days.
* Willing to travel for PET scanning

Exclusion:

* Other major psychiatric disorders such as schizophrenia, schizoaffective illness; current drug or alcohol abuse (within past 2 months), or drug or alcohol dependence <6mos ago; anorexia nervosa or bulimia nervosa in the past year; IV drug use or ecstasy use more than two times.
* A first-degree family history of schizophrenia if the subject is less than 33 years old (mean age of onset for schizophrenia plus two standard deviations).
* Significant active physical illness particularly those that may affect the brain or serotonergic system including blood dyscrasias lymphomas, hypersplenism, endocrinopathies, renal failure or chronic obstructive lung disease, autonomic neuropathies, peripheral vascular disease, diabetes, low hemoglobin and malignancy, significant anemic disease or blood loss and the lab parameters platelet count < 80,000.
* Lacks capacity to consent.
* Actively suicidal-begins expressing a plan for suicide during the washout phase or develop suicidal ideation that warrants admission or requires medication or treatment intervention.
* Electroconvulsive therapy (ECT) within the past 6 months.
* Pregnancy, currently lactating; planning to conceive during the course of study participation or abortion in the past two months.
* Metal implants, pacemaker or metal prostheses or orthodontic appliances, the presence of shrapnel
* Current, past or anticipated exposure to radiation, that may include: being badged for radiation exposure in the workplace, participation in nuclear medicine procedures, including research protocols in the last year.
* A neurological disease or loss of consciousness for more than a few minutes
* Medicinal Patch (participants will be asked to remove before MRI)
* Patients who are responding satisfactorily to psychiatric medications, because they will not be washed-out for purposes of this study
* A documented history of a lack of response to a trial of adequate dose and duration of both lithium and lamotrigine defined as minimal clinical response to lamotrigine 200 mgs for at least 4 weeks or lithium serum levels of at least 0.8 (or dose >= 900 mgs) for at least 4 weeks.
* Patient is unlikely to be able to tolerate medication washout
* Claustrophobia
* Blood donation within 8 weeks of the start of the study.
* History of bleeding disorder or are currently taking anticoagulants.
* Past unsuccessful treatment of Lithium of adequate dose and duration.

HEALTHY CONTROLS

Inclusion:

* No lifetime history of Axis I disorders
* Age range 18-65 years.
* Willing to travel for PET scanning.

Exclusion:

* Past or present alcohol/substance abuse or dependence; IV drug use or ecstasy use more than two times.
* A first-degree relative with history of major depression, schizophrenia, schizoaffective disorder, or suicide attempt; two or more first degree relatives with a history of substance dependence.
* Significant active physical illness particularly those that may affect the brain or serotonergic system including blood dyscrasias lymphomas, hypersplenism, endocrinopathies, renal failure or chronic obstructive lung disease, autonomic neuropathies, peripheral vascular disease, diabetes, low hemoglobin and malignancy, significant anemic disease or blood loss, and the following lab parameters: platelet count < 80,000
* Lacks capacity to consent
* Pregnancy, currently lactating; planning to conceive during the course of study participation or abortion in the past two months
* Metal implants, pacemaker or metal prostheses or orthodontic appliances, the presence of shrapnel
* Current, past or anticipated exposure to radiation, that may include: being badged for radiation exposure in the workplace, participation in nuclear medicine procedures, including research protocols in the last year.
* A neurological disease or loss of consciousness for more than a few minutes
* Medicinal Patch (participants will be asked to remove before MRI)
* Subjects on drugs or medication that affect the serotonin system
* Claustrophobia
* Blood donation within 8 weeks of the start of the study.
* History of bleeding disorder or are currently taking anticoagulants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-11-08 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Parsey, MD, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

REFERENCES:
- [Derived] Ananth M, Bartlett EA, DeLorenzo C, Lin X, Kunkel L, Vadhan NP, Perlman G, Godstrey M, Holzmacher D, Ogden RT, Parsey RV, Huang C. Prediction of lithium treatment response in bipolar depression using 5-HTT and 5-HT1A PET. Eur J Nucl Med Mol Imaging. 2020 Sep;47(10):2417-2428. doi: 10.1007/s00259-020-04681-6. Epub 2020 Feb 13. PMID 32055965

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of Recruitment: 11/2011 - 05/2017 Location: University Medical Centers (Columbia, Stony Brook University)
Pre-assignment Details: 1. Inclusion/Exclusion Criteria must be met prior to beginning study protocols.
  2. Wash-out Period: For participants in the patient group, all were required to be 3 weeks medication free before beginning the study.
Groups:
- Patients With Depression: Patients in this condition will receive lithium administered as follows: Day 1, 2 and 3, 300 mg bid; Days 4-7 lithium 300 qam and 600 qhs. Lithium level will be checked as close to Day 7 as possible and titrated to a therapeutic plasma level of 0.8-1.2 mEq/l. Subjects will not undergo lithium monotherapy if they have a documented history of at least two failed trials of lithium of at least 4 weeks duration with therapeutic blood levels for a major depressive episode
  Lithium
- Healthy Volunteers: Participants in this group underwent baseline assessment for Hamilton Depression Rating Scale and Baseline PET and MRI Imaging. No treatment was provided for this group.
Period: Overall Study
Arm/Group | Patients With Depression | Healthy Volunteers
Started | 47 | 29
Completed | 19 | 29
Not Completed | 28 | 0
Not completed — Diagnosis: Unipolar Depression | 12 | 0
Not completed — Lost to Follow-up | 11 | 0
Not completed — Poor Tolerance to Lithium/Declined Treatment | 5 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants reflected in each group are those that were available for both PET and HDRS-24 baseline measures that also met quality control standards for the imaging data. This number differs slightly from total participants enrolled.
Groups:
- Patients With Depression: Patients with Bipolar depression will receive lithium administered as follows: Day 1, 2 and 3, 300 mg bid; Days 4-7 lithium 300 qam and 600 qhs. Lithium level will be checked as close to Day 7 as possible and titrated to a therapeutic plasma level of 0.8-1.2 mEq/l. Subjects will not undergo lithium monotherapy if they have a documented history of at least two failed trials of lithium of at least 4 weeks duration with therapeutic blood levels for a major depressive episode
  Lithium
- Total: Total of all reporting groups
Arm/Group | Patients With Depression | Healthy Volunteers | Total
Number analyzed (Participants) | 31 | 23 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 23 | 54
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 16 | 11 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 23 | 16 | 39
  Unknown or Not Reported | 6 | 0 | 6
Hamilton Depression Rating Sale [Mean (Standard Deviation); unit: units on a scale] — Patients will have a Hamilton Depression Rating Scale-24 (HDRS) score obtained at baseline. Minimum score 0, maximum possible score 75; the higher the score on the scale, the more severe the degree of depression. Participants must have an HDRS score of at least 15 to be eligible.
  units on a scale | 26.19 (5.86) | 1.62 (2.10) | 16.71 (13.27)

OUTCOME MEASURES:

1. Primary Outcome: Post-Lithium Treatment Hamilton Depression Rating Scale (HDRS)
Description: Patients will have a Hamilton Depression Rating Scale-24 (HDRS) score obtained at baseline. Minimum score 0, maximum possible score 75; the higher the score on the scale, the more severe the degree of depression. Participants must have an HDRS score of at least 15 to be eligible. After eight weeks of medication treatment, the HDRS score will be reevaluated with the HDRS-24 (and rescanned with PET and MRI). Participants who have a 50% or greater decrease in their HDRS-24 score will be considered responders (to Lithium treatment).
Time Frame: 8 weeks
Population: Pre-to-Post lithium treatment change in HDRS Score
Measure: Mean (Standard Deviation); unit: Percent Change in HDRS-24 Score
Groups:
- Patients With BPD: Participants in this group included patients with bipolar depression who were subsequently treated with Lithium. Following baseline PET and MRI scans, treatment was initiated with lithium monotherapy. In brief: days 1-3: 300mg 2x/day, days 4-7: 300mg every morning and 600mg every night; titration to a therapeutic plasma level of 0.8-1.2 mEq/l. Following eight weeks of treatment, patients were rescanned with PET and MRI and reassessed with the HDRS-24.
Arm/Group | Patients With BPD
Number analyzed (Participants) | 19
Percent Change in HDRS-24 Score | -44.49 (34.17)

2. Primary Outcome: Prediction of Treatment Response
Description: Outcome measures were generated following LASSO linear regression analysis using pretreament HDRS-24 AND..
  1. pre-treatment 5-HTT OR
  2. pretreatment 5-HT1A OR
  3. the combination of both 5-HTT and 5-HT1A binding potential
     * to predict post-treatment response defined by a dichotomous remission status variable (remitter vs. non-remitter, where remitter is defined a priori by HDRS-24 <10 post-treatment and a reduction of greater than or equal to 50% in HDRS-24 pre-to-post treatment). Outcome measure is reported as percent accuracy, sensitivity, or specificity in predicting remitter status outcomes.
Time Frame: 8 Weeks
Population: Remission status prediction by groups: accuracy, specificity, and sensitivity. The analyzed population here must have completed both pre- and post-treatment scans for BOTH 5-HTT and 5-HT1A and have 8 weeks of HDRS-24 followup so the predictive power of each individual tracer could be assessed as well as the combination of the two tracers. This is a smaller population that each tracer individually or the outcome of the HDRS-24 scale alone.
Measure: Number; unit: Percentage
Groups:
- Prediction by Pre-treatment 5-HTT: Data analysis to determine whether pre-treatment 5-HTT binding potential along with pre-treatment HDRS-24 predicted treatment response (remission status).
- Prediction by Pre-treatment 5-HT1A: Data analysis to determine whether pre-treatment 5-HT1A binding potential along with pre-treatment HDRS-24 predicted treatment response (remission status).
- Combinatorial Prediction Using Pre-Treatment 5-HTT & 5-HT1A: Data analysis to determine whether pre-treatment 5-HTT & 5-HT1A binding potential along with pre-treatment HDRS-24 predicted treatment response (remission status).
Arm/Group | Prediction by Pre-treatment 5-HTT | Prediction by Pre-treatment 5-HT1A | Combinatorial Prediction Using Pre-Treatment 5-HTT & 5-HT1A
Number analyzed (Participants) | 14 | 14 | 14
Percentage
  Prediction Accuracy = True positive + negative divided by the sum of true + false positive/negative | 71.4 | 85.7 | 84.6
  Prediction Specificity = True negatives divided by the sum of true negative and false positive | 77.8 | 87.5 | 87.5
  Prediction Sensitivity= True positives divided by the sum of true positive and false negative | 60 | 80 | 60

3. Secondary Outcome: Group Differences in 5-HTT Binding Potential
Description: Differences in mean of 5-HTT binding potential between patients with depression pre-treatment, post-treatment, compared to healthy volunteers. Broadly, binding potential is defined as the ratio of the tracer concentration in tissue to the free plasma concentration. It is a measure of the density of "available" targets (e.g. 5-HTT) & the affinity of the ligand (tracer) to that target.
Time Frame: 8 Weeks
Population: Comparison of mean binding potential across patients pre-treatment, post-treatment, and controls.
Measure: Mean (Standard Error); unit: Weighted Mean Binding Potential
Groups:
- Healthy Volunteers: Control participants for baseline measures
- Pre-treatment 5-HTT Binding Potential (Baseline): Participants that presented with Bipolar depression upon enrollment into the study
- Post-treatment 5-HTT Binding Potential (8 Weeks): Participants that presented with Bipolar depression and were treated with Lithium for 8 weeks.
Arm/Group | Healthy Volunteers | Pre-treatment 5-HTT Binding Potential (Baseline) | Post-treatment 5-HTT Binding Potential (8 Weeks)
Number analyzed (Participants) | 23 | 19 | 14
Weighted Mean Binding Potential
  Grey Matter of Cerebellum | 93.27 (17.86) | 88 (1.87) | 88.70 (21.71)
  Midbrain | 264.82 (32.47) | 81.73 (18.59) | 181.13 (90.20)
  Anterior Cingulate | 131.80 (26.99) | 187.48 (60.73) | 130.04 (30.73)
  Amygdala | 198.56 (27.64) | 116.94 (28.73) | 166.73 (61.75)

4. Secondary Outcome: Group Differences in 5-HT1A Binding Potential
Description: Differences in mean of 5-HT1A binding potential between patients with depression pre-treatment, post-treatment, compared to healthy volunteers. Broadly, binding potential is defined as the ratio of the tracer concentration in tissue to the free plasma concentration. It is a measure of the density of "available" targets (e.g. 5-HT1A) & the affinity of the ligand (tracer) to that target.
Time Frame: 8 Weeks
Population: Comparison of mean binding potential across patients pre-treatment, post-treatment, and controls.
Measure: Mean (Standard Error); unit: Weighted Mean Binding Potential
Groups:
- Pre-treatment 5-HT1A Binding Potential (Baseline): Participants that presented with Bipolar depression upon enrollment into the study
- Post-treatment 5-HT1A Binding Potential (8 Weeks): Participants that presented with Bipolar depression and were treated with Lithium for 8 weeks.
Arm/Group | Healthy Volunteers | Pre-treatment 5-HT1A Binding Potential (Baseline) | Post-treatment 5-HT1A Binding Potential (8 Weeks)
Number analyzed (Participants) | 23 | 17 | 13
Weighted Mean Binding Potential
  Raphe Nucleus | 8.91 (3.15) | 9.62 (1.79) | 8.57 (2.58)
  Parahippocampal Gyrus | 12.48 (2.41) | 14.88 (3.13) | 15.79 (3.75)
  Amygdala | 20.8 (5.26) | 17.86 (4.39) | 14.01 (3.41)
  Hippocampus | 27.06 (8.40) | 30.17 (7.84) | 28.39 (7.73)

5. Secondary Outcome: Relationship Between Change in 5-HTT or 5-HT1A Binding Potential Pre- to Post Treatment and Lithium Treatment Response
Description: Linear regression & correlation to assess the relationship between between change in binding potential pre- to post treatment vs. treatment response
Time Frame: 8 weeks
Population: Linear regression between change in PET binding potential pre and post treatment and treatment response.
Measure: Number; unit: Percent Change in Binding Potential
Groups:
- Change in 5-HTT Binding Potential vs. Treatment Response; Change in 5-HT1A Binding Potential and Treatment Response: Data analysis to determine whether there is relationship between the change in 5-HTT binding potential and treatment response.
Arm/Group | Change in 5-HTT Binding Potential vs. Treatment Response | Change in 5-HT1A Binding Potential and Treatment Response
Number analyzed (Participants) | 14 | 13
Percent Change in Binding Potential
  R-Squared: 5-HTT Midbrain | 0.061 | NA — Region not analyzed for this tracer due to lack of target.
  R-Squared: 5-HT1A Raphe | NA — Region not analyzed for this tracer due to lack of target. | 0.086
  R-Squared: 5-HT1A Hippocampus | NA — Region not analyzed for this tracer due to lack of target. | 0.073

ADVERSE EVENTS:
Time Frame: Full study duration for participants: enrollment through final data collection (approximately 6 months)
Description: Definitions for adverse event and/or serious adverse event used to collect adverse event information matches clinicaltrials.gov.
Groups:
- Patients With Depression: Bipolar patients with this condition will receive lithium administered as follows: Day 1, 2 and 3, 300 mg bid; Days 4-7 lithium 300 qam and 600 qhs. Lithium level will be checked as close to Day 7 as possible and titrated to a therapeutic plasma level of 0.8-1.2 mEq/l. Subjects will not undergo lithium monotherapy if they have a documented history of at least two failed trials of lithium of at least 4 weeks duration with therapeutic blood levels for a major depressive episode
  Lithium
Arm/Group | Patients With Depression | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/29
Other Adverse Events (participants affected / at risk) | 0/47 | 0/29

LIMITATIONS AND CAVEATS:
Limitations include: 1. a small sample size, which precludes investigation into interaction factors (e.g. sex/BPD subtype); 2. a short washout duration (3 weeks for ethical reasons), which may not be sufficient to abate treatment effects; 3. scans for both patients and controls conducted across multiple sites, though, importantly, all pre- and post-treatment scans within-participant were conducted at the same site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT01880957/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT01880957/SAP_001.pdf